CLINICAL TRIAL: NCT00006346
Title: Stress Reduction For Breast Cancer in Women 55 Years of Age or Older: Enhancing Quality of Life and Survival
Brief Title: Stress Reduction in Older Women With Stage II, Stage III, or Stage IV Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: SJHCH-TM1; CDR0000068177 (Registry Identifier: PDQ (Physician Data Query)); NCI-V00-1618
Record Dates: First submitted 2000-10-04; First posted 2003-09-04 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2010-03

CONDITIONS: Breast Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; psychosocial effects of cancer and its treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Transcendental meditation may be an effective way to decrease the amount of stress in older women with breast cancer. It is not yet known if transcendental meditation is more effective than basic breast cancer education in improving quality of life.

PURPOSE: This randomized clinical trialstudies stress reduction in improvingquality of life in older women with stage II, stage III, or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effects of active stress reduction with transcendental meditation vs basic breast cancer education on quality of life and survival time in older women with stage II, III, or IV breast cancer.
* Determine behavioral mechanisms that may mediate the effects of stress reduction on survival in these patients.
* Determine baseline variables that contribute to predicting survival time in these patients.

OUTLINE: This is a randomized, single blind (to medical staff), multicenter study. Patients are stratified according to age and participation in support groups. Patients with stage IV disease are also stratified according to type of metastases (visceral vs non-visceral) and timing of metastases (first diagnosis vs recurrence). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive usual medical care and instruction on stress reduction using transcendental meditation (TM), which involves a standard 7-step course. Patients attend training for approximately 1-1.5 hours per session for a total of 6 sessions over 1 week, while receiving usual medical care. Patients then practice TM twice a day for 20 minutes. Patients attend group meetings for approximately 90 minutes once or twice monthly for 6 months to ensure proper technique and understanding.
* Arm II: Patients receive usual medical care and basic literature on breast cancer.

Quality of life is assessed at baseline and then every 6 months for up to 3 years.

Patients are followed monthly for up to 2.5 years.

PROJECTED ACCRUAL: Approximately 166 patients (83 per treatment arm) will be accrued for this study within 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage II, III, or IV breast cancer
* No brain or CNS metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 55 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No non-cancer life-threatening illness
* No history of major psychiatric disorders
* No drug abuse dependency disorder

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhoda S. Pomerantz, MD, MPH, Study Chair — Unity Health Toronto
Locations (3):
- United States (3):
  - St. Joseph Hospital, Chicago, Illinois
  - Hope Center, Terre Haute, Indiana
  - Maharishi International University, Fairfield, Iowa

REFERENCES:
- [Result] Nidich SI, Fields JZ, Rainforth MV, Pomerantz R, Cella D, Kristeller J, Salerno JW, Schneider RH. A randomized controlled trial of the effects of transcendental meditation on quality of life in older breast cancer patients. Integr Cancer Ther. 2009 Sep;8(3):228-34. doi: 10.1177/1534735409343000. PMID 19815592